CLINICAL TRIAL: NCT03249753
Title: to Evaluate the Effect of Food Intake on the Pharmacokinetic of Single Dose SPH3127 Tablets in Chinese Health Subjects
Brief Title: The Effect of Food Intake on the Pharmacokinetic of Single Dose SPH3127 Tablets in Chinese Health Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPH3127-103
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — SPH3127

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPH3127 200mg Panel A (Experimental): Participants who are in panel A will receive a single dose of a SPH3127 tablets 200mg when limosis, then fast 4h after dosing, and 72 hours later participants take the second dose of SPH3127 200mg after a high-fat breakfast.
  Interventions: Drug: SPH3127 200mg Panel A
- SPH3127 200mg Panel B (Experimental): Participants who are in panel B will receive a single dose of a SPH3127 tablets 200mg after a high-fat breakfast, then 72 hours later participants take the second dose of SPH3127 200mg when limosis.
  Interventions: Drug: SPH3127 200mg Panel B

INTERVENTIONS:
Drug: SPH3127 200mg Panel A — Participants who are in panel A will receive a single dose of a SPH3127 tablets 200mg when limosis, then fast 4h after dosing, and 72 hours later participants take the second dose of SPH3127 200mg after a high-fat breakfast.
  Other Names: SPH3127 is a new study drug for hypertension
  Arms: SPH3127 200mg Panel A
Drug: SPH3127 200mg Panel B — Participants who are in panel B will receive a single dose of a SPH3127 tablets 200mg after a high-fat breakfast, then 72 hours later participants take the second dose of SPH3127 200mg when limosis.
  Other Names: SPH3127 is a new study drug for hypertension
  Arms: SPH3127 200mg Panel B

SUMMARY:
This study is a single-center, randomized, open, double-cycle and double-cross and self-reflection phase Ic clinical trial, to evaluate effect and safety of high fat diet on pharmacokinetics of SPH3127 tablets.

Two panels, each consisting of ten participants (The number of single-sex subjects is not less than 1/3 of the total number) will be randomized to A or B groups.

DETAILED DESCRIPTION:
Participants who are in panel A will receive a single dose of a SPH3127 tablets 200mg when limosis, then fast 4h after dosing, and 72 hours later participants take the second dose of SPH3127 200mg after a high-fat breakfast.

Participants who are in panel B will receive a single dose of a SPH3127 tablets 200mg after a high-fat breakfast, then 72 hours later participants take the second dose of SPH3127 200mg when limosis.

ELIGIBILITY:
Inclusion Criteria:

* The body mass index is 19 ~ 26kg/m2 (including the critical value), which allows the minimum weight of male to be 50kg (including the critical value) and 45kg (the critical value) for women.
* Before the study, participants have kown about the significance, potential benefits, inconveniences and potential risks of the study and can follow the research's procedure and already sign the informed consent

Exclusion Criteria:

* Participant who pregnancy, lactating women, and plan to get pregnant within six months after the clinical trial
* Participant who has significant abnormal physical examination, laboratory examination results (such as: liver function examination - aspartate aminotransferase (AST) and alanine aminotransferase (ALT) more than 1.5 times that of the upper limit of normal)
* Participant who has a history of cardiovascular, liver, kidney, digestive tract, nervous system, blood system, familial hematologic disease, abnormal thyroid function, or mental abnormality
* Participant who has drug allergy history, allergy constitution
* Participant who took oral contraceptives within 6 weeks
* Participant who used any drug (including Chinese herbal medicine) within 1 week
* Participant who donated blood within 2 months
* Participant who participated clinical trials of any drug in the past 3 months (as subjects)
* Participant who has any positive result of virus serology check : human immunodeficiency virus antigen antibody (HIV Ag/Ab) and hepatitis c virus (HCV) - Immunoglobulin G（IgG)antibody to IgG, hepatitis b surface antigen (HBsAg) and treponema pallidum antibody (TP)
* Participant who are smoking, drinking, drinking coffee, strong tea and drug abusers
* Participant who the researchers believe that there are volunteers who are not suitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-23 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Plasma area under curve（AUC）(0-∞) of SPH3127 3127 | Before dose, and at 0.17 hours、0.33h、0.5h、0.75h、1h、1.25h、1.5h、2h、4h、6h、8h、12h、24h hours after dose
  to evaluate the area under curve（AUC）(0-∞) of SPH3127 by feeding
Plasma Cmax of SPH3127 | Before dose, and at 0.17 hours、0.33h、0.5h、0.75h、1h、1.25h、1.5h、2h、4h、6h、8h、12h、24h hours after dose
  to evaluate the Cmax of SPH3127 by feeding
Plasma Tmax of SPH3127 | Before dose, and at 0.17 hours、0.33h、0.5h、0.75h、1h、1.25h、1.5h、2h、4h、6h、8h、12h、24h hours after dose
  to evaluate the Tmax of SPH3127 by feeding
Apparent terminal half-life of SPH3127 | Before dose, and at 0.17 hours、0.33h、0.5h、0.75h、1h、1.25h、1.5h、2h、4h、6h、8h、12h、24h hours after dose
  to evaluate the Apparent terminal half-life of SPH3127 by feeding

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Baseline to 10-13 days post last dose
  Incidence and intensity of Adverse Events according to Common Toxicity Criteria (CTC version 4.03) associated with SPH3127
Change from baseline in laboratory hematology values | Baseline to 10-13 days post last dose
  to evaluate the change from baseline in laboratory hematology values
Change from baseline in laboratory chemistry values | Baseline to 10-13 days post last dose
  to evaluate the Change from baseline in laboratory chemistry values
Change from baseline in ECG | Baseline to 10-13 days post last dose
  to evaluate the from baseline in ECG

CONTACTS AND LOCATIONS:
Locations (1):
- The capital medical university affiliated Beijing anzhen hospital, Beijing, Beijing Municipality, China